CLINICAL TRIAL: NCT06324708
Title: Finite-element Analysis Based on Computed Bone Mineralometry (DXA) as an Aid to Pre and Post Assessment in Hip Arthroplasty Surgery
Brief Title: Analysis of Defined Elements on DXA in Patients Undergoing Hip Arthroplasty
Acronym: THA_DXA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: THA_DXA
Record Dates: First submitted 2024-01-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-01

CONDITIONS: Bone Resorption; Arthroplasty Complications
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip arthroplasty group (Experimental): This single group is composed by patients undergoing hip arthroplasty
  Interventions: Diagnostic Test: DXA

INTERVENTIONS:
Diagnostic Test: DXA — Patients will undergo a femoral and lumbar DXA

SUMMARY:
The purpose of this study is to investigate the role of two-dimensional FEM models obtained from DXA images in the longitudinal assessment of periprosthetic bone, in subjects undergoing hip arthroplasty. Specifically, the study will focus on the joint analysis of changes in the parameters of bone mineral density (BMD) and Bone Strain Index (BSI) at the level of periprosthetic bone of the proximal femur in patients undergoing hip replacement surgery using DXA, evaluating the densitometric variation of these two parameters over time, starting from an immediately postoperative data and checking the change at 6 months to follow the patient through the postoperative course

DETAILED DESCRIPTION:
Hip osteoarthritis is nowadays one of the most prevalent diseases in developed countries. Prosthetic replacement of the degenerated joint is the definitive treatment for more advanced stages of osteoarthritis.

Despite continuous improvements in prosthesis material, design, and implantation procedures that have led to a percentage reduction in failures, there is still an albeit low risk of hip prosthetic implantation failure today.

Preoperative planning is therefore a prerequisite in order to ensure the success of the implant and its longterm survival. This is generally based on radiographic investigations, with implant selection being based on "templating" the radiographs to replicate the patient's joint anatomy.

However, with preoperative radiographs (or possibly second-level investigations such as CT scans), only the geometry of the bone subjected to the implant through is evaluated, without obtaining information regarding the bone density or the load to which the implant will be subjected. However, the long-term stability of the implant depends on the load transfer to the adjacent bone. Non-physiological load transfer can cause stress-shielding, bone resorption, or fibrous tissue growth due to high micromovements at the implant-bone interface.

The study of images by finite element analysis (FEA) has been used in orthopedic biomechanics for fifty years, and the techniques have progressively evolved in terms of sophistication and ability to assess the postoperative mechanical environment The Bone Strain Index (BSI) software, obtained from computerized bone mineral imaging (DXA) surveys using FEA, automatically calculates the deformations and stresses to which a given bone segment is subjected from patient-specific loading conditions. Previous studies have evaluated changes in periprosthetic bone mineral density (BMD) around hip replacement, noting densitometric changes that could vary between subjects and as a function of treatment, suggesting periprosthetic DXA as a useful technique in early assessment of possible bone loss from periprosthetic resorption. However, there are no DXA-based studies in the literature that correlate BMD changes to periprosthetic mechanical stress.

In this study, the investigators aim to study periprosthetic hip bone by DXA technique, applying the FEA method to obtain two-dimensional models of bone resistance to loading, using BSI software.

This evaluation will be included in the context of the normal pre- and postoperative evaluation process, with a view to better understanding the therapeutic outcome and possibly providing a means of predicting early mobilization and thus possible surgical failure.

Patients will be recruited as part of the normal surgical procedure for patients referred for hip replacement surgery to be performed at the Galeazzi - Sant'Ambrogio Hospital. Subjects, after being informed about the study and giving their written informed consent, will provide the examining physician with the information needed to fill out appropriate biographical and medical history forms. Recruitment will be entrusted to the physicians who will perform routine clinical examinations.

Once enrolled, patients will have a lumbar and femoral DXA scan as a preoperative preliminary investigation; anthropometric evaluations, postoperative DXA scans (immediate postoperative and at 3,6,12 months), blood draws, and PROMs will be administered for each patient. The study will be conducted according to the guidelines of Good Clinical Practices

ELIGIBILITY:
Inclusion Criteria:

Patients who are candidates for elective hip arthroplasty surgery (indication determined only by the Orthopedic Surgeon)

* Patients with noninflammatory degenerative hip joint disease, including osteoarthritis and the outcomes of congenital hip dysplasia.
* Hip joint deformity correction surgery
* Patients aged 50 to 90 years (completed)
* 18 ≤ Body Mass Index (BMI) ≤ 35 kg/m2
* Postmenopausal women (absence of menstrual cycle for at least 2 years)
* Willingness and ability to provide informed consent

Exclusion Criteria:

Taking drugs that may interfere with muscle or bone metabolism,

* Evidence of diseases known to interfere with bone or muscle metabolism
* Rheumatoid arthritis
* Patients undergoing revision hip replacement surgery
* Presence of infection or suspicion of infection at the hip
* Inability to provide informed consent
* Previous synthetic surgery for proximal femur fractures
* Severe obesity (BMI >35kg/m2)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Role of two-dimensional FEM models obtained from DXA images in longitudinal evaluation of periprosthetic bone | 12 months
  The purpose of this study is to investigate the role of two-dimensional FEM models obtained from DXA images in longitudinal evaluation of periprosthetic bone, in subjects undergoing hip arthroplasty.
  Specifically, the study will focus on the joint analysis of changes in the parameters of bone mineral density (BMD) [g/cm2] and Bone Strain Index (BSI) at the periprosthetic bone level of the proximal femur in patients undergoing hip implant surgery using DXA, evaluating the densitometric change of these two parameters over time, starting from an immediately postoperative data and verifying the change at 6 months, to follow the patient through the postoperative course. Since there are no longitudinal evaluation studies of periprosthetic stress, measured by finite element analysis with BSI software, it was decided to focus on the variations in BMD as the main result, limiting the observation on the behavior of the BSI parameter with respect to the variations in BMD.

SECONDARY OUTCOMES:
Role of two-dimensional FEM models of bone resistance to loading | 12 months
  To investigate the role of two-dimensional FEM models of bone resistance to loading, obtained from DXA scans using BSI software in various femoral and acetabular periprosthetic regions.
Identification of mechanical stress | 12 months
  To identify, by joint assessment of BMD and BSI, which periprosthetic regions are most subjected to mechanical stress by virtue of the presence of the prosthesis, in order to predict possible excessive periprosthetic bone resorption
Assesment with PROMs: VAS | 12 months
  Assessment of patients' health status through the collection of visual analogue scale (VAS). Will be used a linear scale with no pain at the left border and very serious pain at the right border
Assesment with PROMs; HHS | 12 months
  Assessment of patients' health status through the collection of Harris Hip Score (HHS). The score is composed by question with multiple choice. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Assesment with PROMs: SF12 | 12 months
  Assessment of patients' health status through the collection of SF12. The SF-12 is made up of 4 scales (physical functioning, role and physical health, role and emotional state, mental health) measured by 2 items each and 4 scales each measured by one item (physical pain, vitality, social activities and general health).
Assesment with PROMs: HOOS PS | 12 months
  Assessment of patients' health status through the collection of Hip Disability and Osteoarthritis Outcome Score (HOOS PS). The questionnaire includes just 5 items with 5 response options each. Only one answer can be selected. Each of the items is scored from 0 (no health problems) to 4 (severe health problems). A raw score is generated by summing up all points of the 5 answers (maximum raw score = 20).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mangiavini, Principal Investigator — University of Milan, IRCCS Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy

IPD SHARING:
Plan to Share IPD: No